CLINICAL TRIAL: NCT07171385
Title: Persistent Neuromuscular Deficits in the Posterior Kinetic Chain Following Hamstring Strain Injury: A Cross-Sectional Study Using EMG
Brief Title: Posterior Chain EMG Patterns in Athletes With and Without Hamstring Injury
Status: Completed | Type: Observational
Sponsor: Ankara Yildirim Beyazıt University (Other)
Collaborators: Mersin University (Other); T.C. Dumlupınar Üniversitesi (Other); Eskisehir Technical University (Other); Istanbul Gelisim University (Other); Çanakkale Onsekiz Mart University (Other); Saglik Bilimleri Universitesi (Other); Manisa Celal Bayar University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-350
Record Dates: First submitted 2025-09-06; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Muscle Strain; Neuromuscular Diseases; Athletic Injuries
Keywords: Hamstring Muscles; Electromyography; Athletic Injuries; Muscle, Skeletal; Exercise Therapy; Soccer; Rehabilitation; Biceps Femoris; Nordic Hamstring Curl; Kettlebell Swing; Supine Sliding Leg Curl; Reinjury Prevention
MeSH Terms: conditions — Sprains and Strains; Neuromuscular Diseases; Athletic Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Injured Group: Male football players aged 18-30 years with a history of unilateral hamstring strain injury (HSI) within the past 6 months, BMI 18.5-24.9 kg/m², able to perform study exercises (Nordic Hamstring Curl, Kettlebell Swing, Supine Sliding Leg Curl). Surface electromyography (sEMG) was used to measure activation of biceps femoris, gluteus maximus, latissimus dorsi, and iliocostalis lumborum during a single session. No interventions were applied (observational study).
  Interventions: Other: Nordic Hamstring Curl (NHC); Other: Kettlebell Swing (KS); Other: Supine Sliding Single-Leg Curl (SSLC)
- Healthy Control Group: Male football players aged 18-28 years, no history of hamstring strain injury in the past 6 months, BMI 18.5-24.9 kg/m², straight-leg raise on dominant limb <80°, able to perform study exercises (Nordic Hamstring Curl, Kettlebell Swing, Supine Sliding Leg Curl). Surface electromyography (sEMG) measured activation of biceps femoris, gluteus maximus, latissimus dorsi, and iliocostalis lumborum in a single session. No interventions were applied (observational study).
  Interventions: Other: Nordic Hamstring Curl (NHC); Other: Kettlebell Swing (KS); Other: Supine Sliding Single-Leg Curl (SSLC)

INTERVENTIONS:
Other: Nordic Hamstring Curl (NHC) — Knee-dominant eccentric hamstring strengthening exercise performed on a padded surface. Participants control the descent of the torso while knees remain fixed, emphasizing eccentric activation of hamstring muscles.
Other: Kettlebell Swing (KS) — Hip-dominant ballistic movement involving rapid hip flexion-extension using a kettlebell (16-20 kg depending on participant's ability). Each repetition includes concentric, isometric, and eccentric phases standardized by metronome pacing.
Other: Supine Sliding Single-Leg Curl (SSLC) — Closed-chain exercise performed in supine position with heels placed on sliding discs. One leg is extended while the other leg performs concentric-eccentric sliding curl.

SUMMARY:
This cross-sectional observational study investigated posterior chain muscle activation patterns in football players with and without a history of hamstring strain injury. Forty-two male athletes were assessed using surface electromyography (sEMG) during Nordic Hamstring Curl, Kettlebell Swing, and Supine Sliding Leg Curl exercises. Results demonstrated persistent deficits in biceps femoris, gluteus maximus, latissimus dorsi, and iliocostalis lumborum activation in previously injured athletes compared to controls, suggesting that neuromuscular alterations extend beyond the hamstring itself and may increase reinjury risk.

ELIGIBILITY:
Inclusion Criteria:

* Male football players, aged 18-30 years
* Body mass index (BMI) between 18.5-24.9 kg/m²
* Voluntary participation and written informed consent
* Ability to perform all test exercises (Nordic Hamstring Curl, Kettlebell Swing, Supine Sliding Single-Leg Curl)
* For injured group: unilateral hamstring strain within the past 6 months
* For control group: no hamstring injury within the past 6 months

Exclusion Criteria:

* Professional sports background
* Lower or upper extremity injury within the last year (other than index hamstring strain for the injured group)
* Neurological, musculoskeletal, respiratory, or cardiovascular conditions limiting participation
* Recent spinal surgery
* Acute low-back or lower-limb pain
* Sensory impairments interfering with performance
* History of malignancy

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Forty-two male football players aged 18-30 years participated, including 21 with a history of unilateral hamstring strain injury and 21 healthy controls. All were recreational to semi-professional athletes with BMI within the normal range and able to complete functional posterior chain exercises.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2023-11-11 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Gluteus Maximus Activation (%MVIC) | Single laboratory visit; measurements during 3 repetitions of each exercise (Nordic Hamstring Curl, Kettlebell Swing, Supine Sliding Single-Leg Curl)
  Surface EMG amplitude (RMS) normalized to MVIC, averaged across three functional exercises. Mean %MVIC compared between groups.
Biceps Femoris Long Head Activation (%MVIC) | Single laboratory visit; measurements during 3 repetitions of each exercise (Nordic Hamstring Curl, Kettlebell Swing, Supine Sliding Single-Leg Curl)
  Surface EMG amplitude (RMS) normalized to MVIC. Mean %MVIC across repetitions compared between injured and healthy athletes.
Latissimus Dorsi Activation (%MVIC) | Single laboratory visit; measurements during 3 repetitions of each exercise (Nordic Hamstring Curl, Kettlebell Swing, Supine Sliding Single-Leg Curl)
  Surface EMG amplitude (RMS) normalized to MVIC, averaged across three functional exercises. Mean %MVIC compared between groups.
Iliocostalis Lumborum Activation (%MVIC) | Single laboratory visit; measurements during 3 repetitions of each exercise (Nordic Hamstring Curl, Kettlebell Swing, Supine Sliding Single-Leg Curl)
  Surface EMG amplitude (RMS) normalized to MVIC. Mean %MVIC across repetitions compared between injured and healthy athletes.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in this article (text, tables, figures) will be made available upon reasonable request to the corresponding author, following publication. Data will be shared with qualified researchers for academic purposes, subject to ethical approval and institutional data protection policies. Supporting documents (study protocol, statistical analysis plan) may also be provided on request.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified individual participant data (IPD), study protocol, and statistical analysis plan will be available beginning 6 months after publication of the main results article and will remain available for a period of 5 years thereafter.
Access Criteria: Qualified researchers affiliated with academic or research institutions may request access to de-identified IPD, the study protocol, and the statistical analysis plan. Requests must be made in writing to the corresponding author and will be reviewed by the study team. Access will be granted for scientifically sound proposals, with data shared via secure transfer following institutional data protection policies.
URL: https://orcid.org/0000-0002-1524-6295

REFERENCES:
- [Derived] Gulgosteren E, Yuksel O, Gurol B, Yildirim O, Atar O, Soylu C, Altundag E, Acar G. Persistent neuromuscular deficits in the posterior kinetic chain following hamstring strain injury: EMG insights from nordic hamstring curl, kettlebell swing, and supine sliding leg curl. BMC Sports Sci Med Rehabil. 2025 Nov 29;18(1):6. doi: 10.1186/s13102-025-01435-5. PMID 41318473